CLINICAL TRIAL: NCT07117877
Title: Etoposide Capsules Combined With Bevacizumab and Iparomlimab and Tuvonralimab in the Treatment of Platinum Resistant or Platinum Refractory Ovarian Cancer: a Single Arm, Open, Single Center, Phase II Clinical Study
Brief Title: Etoposide Capsules Combined With Bevacizumab and Iparomlimab and Tuvonralimab in the Treatment of Platinum Resistant or Platinum Refractory Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaohua Wu MD [zzhong], Professor, Director of Gynecologic Oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCR-EBQ-2025
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Platinum Resistant Ovarian Cancer; Platinum Refractory Epithelial Ovarian Cancer; Ovarian Cancer (OvCa)
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Etoposide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Etoposide+Bevacizumab+Iparomlimab and Tuvonralimab (Experimental): Participants will receive Etoposide Capsules, Bevacizumab and Iparomlimab and Tuvonralimab in combination. 21 days as a cycle.
  Interventions: Drug: Etoposide Capsules; Drug: Bevacizumab; Drug: Iparomlimab and Tuvonralimab (QL1706)

INTERVENTIONS:
Drug: Etoposide Capsules — 50 mg(25mg/pill, 2 pills at a time) orally, qd, days 1 to 14, per cycle
Drug: Bevacizumab — 7.5mg/kg, i.v, q3w
Drug: Iparomlimab and Tuvonralimab (QL1706) — 5mg/kg, i.v., q3w

SUMMARY:
This study is a Prospective, Single-arm, Phase II clinical trial. The purpose of this study is to find out if taking Etoposide Capsules combined With Bevacizumab and Iparomlimab and Tuvonralimab is safe and works well for people with platinum-resistant or platinum refractory ovarian cancer . Researchers will look at the Progression-Free Survival, Objective Response Rate, Overall Survival, safety, and any side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75, female;
2. According to RECIST 1.1 criteria, there are measurable lesions at baseline;
3. ECOG PS： 0-1；
4. Epithelial ovarian, fallopian tube, and primary peritoneal cancer with platinum resistance or platinum refractory recurrence; Provide 10 white films for pathological type confirmation and efficacy marker exploration, and meet all of the following conditions.

   ① Received systemic treatment with ≥ 1 line and ≤ 6 lines, among which only received systemic treatment with ≤ 4 lines after platinum resistance relapse.

   ② Previous treatments should include at least one platinum based chemotherapy regimen. There are two specific situations:
   1. For patients who have only received 1-line platinum based chemotherapy in the past, disease remission (CR or PR) must be achieved, and disease progression must occur within a period of ≥ 4 weeks and<6 months after the last platinum based chemotherapy.
   2. For patients who have received systemic treatment from line 2 to line 5 in the past, it is required that disease progression must occur within a period of less than 6 months after the last platinum based chemotherapy.

   Note: When determining the number of lines, the following requirements should be noted:

   The overall count of neoadjuvant ± adjuvant systemic therapy is one line. Maintenance treatment does not calculate the number of lines separately. Simple endocrine therapy is counted as a baseline, but the use of endocrine therapy due to non disease progression (such as only elevated CA-125) is not counted as a baseline.

   Changing the treatment plan due to intolerance without disease progression is not considered as changing the line.

   The subject needs to experience disease progression after the final systemic treatment.
5. The main organ functions well and meets the following criteria:

   1. Blood routine examination (without blood transfusion or correction with hematopoietic stimulating factor drugs within 14 days): hemoglobin (Hb) ≥ 90g/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; platelet count (PLT) ≥ 90 × 109/L;
   2. Biochemical examination: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (≤ 5 × ULN for tumor liver metastases); Serum total bilirubin (TBIL) ≤ 1.5 × ULN (Gilbert syndrome subjects, ≤ 3 × ULN); Serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance rate ≥ 60mL/min;
   3. Coagulation function: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5 × ULN;
   4. Urine routine examination shows urinary protein<2+; If urinary protein is ≥ 2+, 24-hour urinary protein quantification should be<1 g;
   5. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ 50%.
6. Non surgical sterilization or female patients of childbearing age are required to use two medically approved contraceptive measures (such as intrauterine devices, birth control pills, or condoms) during the study treatment period and within 3 months after the end of the study treatment period; Female patients of childbearing age who undergo non-surgical sterilization must have a negative serum HCG test within 72 hours before their first medication and must be non lactating; For male patients whose partners are women of childbearing age, two effective methods of contraception should be used during the study treatment period and within 3 months after the end of the study treatment period.
7. The subjects voluntarily joined this study, signed informed consent forms, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Patients who participate in other clinical trials simultaneously;
2. Allergic constitution, including a history of severe drug allergies or drug allergic reactions; Known to be allergic or intolerant to the investigational drug;
3. No measurable lesions or lesions that cannot be evaluated;
4. Patients with untreated central nervous system metastases, who have previously received systemic or curative treatment for brain or meningeal metastases (radiotherapy or surgery), have been confirmed stable for at least one month by imaging, and have stopped systemic hormone therapy (dose>10mg/day prednisone or other therapeutic hormones) for more than two weeks without clinical symptoms can be included;
5. Those who are unable to swallow pills normally or have gastrointestinal dysfunction, as determined by researchers, may affect drug absorption;
6. Individuals who have experienced intestinal obstruction within the past 3 months;
7. At present, there are uncontrollable malignant pleural effusion, ascites, or pericardial effusion (defined as those that cannot be effectively controlled by diuretics or puncture methods as determined by researchers);
8. Suffering from uncontrolled comorbidities, including but not limited to: active HBV or HCV infection; Known history of HIV infection or AIDS; Active syphilis; Active tuberculosis; Active infection; Uncontrolled hypertension and symptomatic heart failure; Active bleeding;
9. History of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or other malignant tumors within 5 years prior to the initial administration of the study (excluding completely relieved carcinoma in situ and malignant tumors with slow progression determined by the investigator)
10. Other incurable malignant tumors in the past (within 5 years) or at the same time, except for cured skin basal cell carcinoma, cervical carcinoma in situ and breast cancer with no recurrence after radical surgery>3 years;
11. Pregnant or lactating women;
12. According to the researchers' assessment, there may be other factors that could lead to the forced termination of this study, such as other serious illnesses (including mental illnesses) requiring concurrent treatment, serious laboratory abnormalities, and family or social factors that could affect the safety of the subjects or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
PFS | approximately 2 years
  Progression-free survival, according to RECIST v1.1

SECONDARY OUTCOMES:
ORR | Up to 24 months
  Objective response rate, according to RECIST v1.1
OS | Up to 2 years
  Overall survival, according to RECIST v1.1
AEs | From the first drug administration to within 30 days for the last treatment dose
  Adverse Events, according to CTCAE V5.0 criteria, During the trial, the adverse event record form should be truthfully filled in, including the occurrence time, severity, correlation with study treatment, duration, measures taken and outcome of the adverse event.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Data is available per require after approved by ethics broad